CLINICAL TRIAL: NCT03403855
Title: Evaluation of Short and Long External Length Rocket® Pleural Catheters in Terms of Quality of Life, Feasibility and Satisfaction in Patients Being Treated for Recurrent Malignant Pleural Effusions
Brief Title: Rocket® Pleural Catheters: QOL, Feasibility and Satisfaction in Recurrent MPE Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20170753-01H
Record Dates: First submitted 2017-10-31; First posted 2018-01-19 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Intervention Model Description: All patients will have a regular full length Rocket catheter inserted at baseline, with an external length of 16cm. All patients will have their catheter length modified at 2 weeks in clinic and shortened to an external length of 5cm. Patient satisfaction will be collected at 2 weeks prior to the modification, and 4 weeks when the patient has a shorter catheter.
  The modification is easily done without any use of anesthesia as it is external to the patient. It is done with the tool kit that comes along with the catheter.
  All patients will be referred to palliative home care services for assistance with drainage. Drainage catheters are usually provided by Ontario Medical Supplies. However, the drainage catheters to be used in this study will be those supplied by Rocket Medical Inc., as they will be providing Dr. Amjadi with some samples to evaluate their product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rocket® IPC- Long External Length (Experimental): Intervention Rocket® IPC- Long External Length: a regular full length (long catheter) Rocket catheter inserted at baseline, with an external length of 16cm. Catheter length will be modified at 2 weeks in clinic, shortened to an external length of 5cm (short catheter). Patient satisfaction will be collected at 2 weeks prior to the modification, and at 4 weeks when the patient has a shorter catheter.
  The modification is easily done without any use of anesthesia as it is external to the patient using the tool kit that comes along with the catheter.
  Patients will be referred to palliative home care services for assistance with drainage. The drainage catheters to be used in this study will be samples supplied by Rocket Medical Inc., for Dr. Amjadi to evaluate their product.
  Interventions: Device: Rocket® IPC- Long External Length
- Rocket® IPC- Short External Length (Experimental): Intervention Rocket® IPC- Short External Length : a regular full length (long catheter) Rocket catheter inserted at baseline, with an external length of 16cm. Catheter length will be modified at 2 weeks in clinic, shortened to an external length of 5cm (short catheter). Patient satisfaction will be collected at 2 weeks prior to the modification, and at 4 weeks when the patient has a shorter catheter.
  The modification is easily done without any use of anesthesia as it is external to the patient using the tool kit that comes along with the catheter.
  Patients will be referred to palliative home care services for assistance with drainage. The drainage catheters to be used in this study will be samples supplied by Rocket Medical Inc., for Dr. Amjadi to evaluate Rocket's product.
  Interventions: Device: Rocket® IPC- Short External Length

INTERVENTIONS:
Device: Rocket® IPC- Long External Length — Rocket® IPC- Long External Length Intervention. Evaluation of Long and Short External Length Rocket® Pleural Catheters in Terms of Quality of Life, Feasibility and Satisfaction in Patients Being Treated for Recurrent Malignant Pleural Effusions
  Arms: Rocket® IPC- Long External Length
Device: Rocket® IPC- Short External Length — Rocket® IPC- Short External Length Intervention. Evaluation of Long and Short External Length Rocket® Pleural Catheters in Terms of Quality of Life, Feasibility and Satisfaction in Patients Being Treated for Recurrent Malignant Pleural Effusions
  Arms: Rocket® IPC- Short External Length

SUMMARY:
This study will take place in Ottawa, Ontario, and will include 100 patients who are receiving tunnelled pleural catheters to treat their symptoms of MPE. The aim of this study is to evaluate the effectiveness of the shorter versus longer external length Rocket® pleural catheter in managing malignant pleural effusions in terms of patients' self-rated quality of life, its ease of use, the incidence of complications, and levels of health care provider satisfaction.

DETAILED DESCRIPTION:
Pleural effusion is a medical condition, which occurs when too much fluid collects in the space between the lungs and the chest wall. This extra fluid makes it hard for the lungs to fully expand and take in enough air when inhaling. Malignant pleural effusions (MPE) are effusions related to cancer. Common symptoms of MPE include: dyspnea (shortness of breath), cough, weight loss, and chest pain. Tunneled pleural catheters (which are inserted into the body) are now commonly used to treat the symptoms of malignant pleural effusions by draining this extra fluid on a daily basis. This drainage can be done and home and need not be performed at a hospital.

The aim of this study is to evaluate the effectiveness of the shorter versus longer external length Rocket® pleural catheter in managing malignant pleural effusions in terms of patients' self-rated quality of life, its ease of use, the incidence of complications, and levels of health care provider satisfaction. The Rocket® pleural catheter has been approved by the Food and Drug Administration (FDA) and Health Canada for the management of malignant pleural effusions.

This study will take place in Ottawa, Ontario, and will include 100 patients who are receiving tunnelled pleural catheters to treat their symptoms of MPE. All information required to evaluate the Rocket® catheter will be collected from routine medical follow-up visits. The period of time for the study is approximately 4 weeks (28 days).

The Rocket® catheter will be provided to patients who wish to participate in this study. If patients do not wish to participate, they will receive the current standard of care (the PleurX catheter) and will undergo the same standard medical assessments that will be performed in this study.

All patients eligible for the study will have a regular full length Rocket catheter inserted at baseline, with an external length of 16cm. All patients will have their catheter length modified at 2 weeks in clinic and shortened to an external length of 5cm.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of symptomatic (BDI < 6), and moderate sized (> 1/3 of hemithorax) MPE
2. Persistent malignant pleural effusion that is free flowing
3. Life expectancy of at least 2 months (approximate duration of follow-up for the study)
4. Age greater than 18
5. Consent to undergoing TPC treatment for recurrent MPE

Exclusion Criteria:

1. Prior attempted chemical pleurodesis on ipsilateral side
2. Active pleural or pulmonary infection
3. Currently hospitalized for reasons other than MPE or in hospice care
4. Life expectancy estimated at less than 2 months
5. Inability to complete questionnaires (English or French)
6. Refusal to give informed consent
7. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients' self-rated quality of life - change from baseline compared to 2 and 4 weeks post catheter insertion. | Assessed at baseline compared to changes at 2 weeks and 4 weeks post catheter insertion. Questionnaires will be administered at routine medical visits on day O, 14, and 28.
  Self-rated QOL at baseline compared to 2 weeks and 4 weeks post catheter insertion.
  Quality of life will be assessed using the validated EORTC QLQ-C30 (European Organization of Research and Treatment of Cancer Quality of Life Evaluation) questionnaire.
Patients' self-rated quality of life on domains specific to lung cancer-change from baseline compared to 2 and 4 weeks post catheter insertion. | Assessed at baseline compared to changes at 2 weeks and 4 weeks post catheter insertion. Questionnaires will be administered at routine medical visits on day O, 14, and 28.
  Self-rated QOL in domains specific to lung cancer will be assessed at baseline compared to 2 weeks and 4 weeks post catheter insertion.
  Quality of life will be assessed using the validated lung cancer specific EORTC QLQ-LC13 (European Organization of Research and Treatment of Cancer (EORTC) Quality of Life QLQ-LC13 disease specific) questionnaire.

SECONDARY OUTCOMES:
Ease of use of the short versus long Rocket® pleural catheter. | Questionnaire will be administered at routine medical visits on day O, 14, and 28.
  Ease of use of the short versus long Rocket pleural catheter as reported by the study doctor as well as the hospital and home care nursing staff.
  Ease of use will be measured using a non-validated questionnaire, which will assess the functionality of the short versus long Rocket® pleural catheter.
Feasibility: measured by incidence of complications (adverse events reports) | Complications will be quantified and described based on patients' reporting of adverse events (at 2 week and 4 week medical assessments). Satisfaction with device questionnaires will be administered at routine medical visits on day 0, 14 and 28.
  Feasibility will be measured by the incidence of complications found in patients using short versus long Rocket® pleural catheters to treat symptoms of MPE as well as hospital and home care nursing staffs' level of satisfaction with the Rocket® catheter.
  The time to removal of the Rocket catheter will also be followed and complications will be quantified and described based on patients' reporting of adverse events (at 2 week and 4 week medical assessments) and ongoing reports from home care nurses. All complications will be documented, the most clinically relevant include pleural infection and cellulitis, pain, and catheter obstruction and symptomatic loculated effusion.

OTHER OUTCOMES:
Levels of Satisfaction with the device | Satisfaction with device questionnaires will be administered at routine medical visits on day 0, 14 and 28.
  Levels of satisfaction with the Rocket® catheter will be measured using a non-validated questionnaire which will assess comfort with the short versus long Rocket® pleural catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Kayvan Amjadi, MD, Principal Investigator — Director Interventional Pulmonology, TOH (General Campus)
Locations (1):
- Ottawa Hospital, General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.